CLINICAL TRIAL: NCT07132996
Title: Correlation of Spleen Size and Hematoma Volume With Clinical Course and 45- Day Mortality in Emergency Patients With Hemorrhagic Stroke
Brief Title: Spleen Volume Change Predicts 45-Day Mortality in Neurocritical Care: A Prospective Cohort Study
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cagdas Yildirim, MD, Assistant Professor, Ankara City Hospital Bilkent
Other Study IDs: E1:24:29; E1 24 29 (Registry Identifier: The Ministry of Health Ankara Bilkent City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Intracerebral Hemorrhage (ICH); Hemorrhagic Stroke, Intracerebral; Neurocritical Care; Acute Brain Injury; Ultrasound
Keywords: spleen volume change; ΔSpleen; ΔHematoma; 45-day mortality risk; neurocritical care
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decreased Spleen Volume Group (ΔSpleen < 0 mL): Patients with spontaneous intracerebral hemorrhage who demonstrated a reduction in splenic volume from baseline to 72 hours after admission (negative ΔSpleen). Outcomes include 45-day all-cause mortality, changes in Glasgow Coma Scale, and inflammatory biomarker levels.
  Interventions: Diagnostic Test: POCUS-based Splenic Volume Measurement
- Stable/ Increased Spleen Volume Group (ΔSpleen ≥ 0 mL): Patients with spontaneous intracerebral hemorrhage who showed no change or an increase in splenic volume from baseline to 72 hours after admission (ΔSpleen ≥ 0 mL). Outcomes include 45-day all-cause mortality, changes in Glasgow Coma Scale, and inflammatory biomarker levels.
  Interventions: Diagnostic Test: POCUS-based Splenic Volume Measurement

INTERVENTIONS:
Diagnostic Test: POCUS-based Splenic Volume Measurement — Splenic volume was measured at baseline and at 72 hours using the Butterfly iQ+ handheld ultrasound (Butterfly Network, Inc.) in abdominal preset mode. Certified POCUS operators obtained spleen length, width, and depth in standard orthogonal planes. Volumes were calculated using the prolate ellipsoid formula (length × width × depth × 0.523), a validated method in ultrasound volumetric studies. ΔSpleen was defined as the 72-hour value minus the baseline value.

SUMMARY:
This study investigates whether changes in spleen size over 72 hours can help predict the risk of death within 45 days in patients who were admitted to the emergency department with a type of bleeding in the brain called intracerebral hemorrhage. The spleen is a key immune organ that may shrink or enlarge in response to injury. A total of 42 adult patients with confirmed intracerebral hemorrhage were enrolled between March and September 2024 at Ankara Bilkent City Hospital in Turkey. Spleen size and brain bleeding volume were measured by imaging tests at the time of admission and repeated 72 hours later. Patients were followed for 45 days to determine survival status. The main goal of the study was to see if spleen size change (ΔSpleen) is a better predictor of death than brain bleeding volume change (ΔHematoma).

DETAILED DESCRIPTION:
This is a prospective observational cohort study designed to evaluate the prognostic value of spleen volume changes in patients with non-traumatic intraparenchymal hemorrhage (ICH). The study was conducted at Ankara Bilkent City Hospital Emergency Department, a tertiary care center with neurocritical care expertise, between March 15, 2024, and September 15, 2024.

A total of 42 consecutive adult patients with neuroimaging-confirmed ICH were enrolled upon admission to the emergency department. All participants underwent baseline brain computed tomography (CT) and abdominal ultrasound within the first hours of presentation. Repeat imaging studies, including brain CT and abdominal ultrasound, were performed at 72 hours after enrollment.

Spleen volume (mL) and hematoma volume (mL) were measured using standardized volumetric methods. The change in each parameter (ΔSpleen and ΔHematoma) was calculated by subtracting the baseline measurement from the 72-hour measurement. Clinical and demographic characteristics, comorbidities, and imaging findings were prospectively collected for each participant.

The primary study objective is to determine whether changes in spleen volume (ΔSpleen) are independently associated with 45-day all-cause mortality in patients with ICH. A secondary objective is to compare the prognostic performance of ΔSpleen with changes in hematoma volume (ΔHematoma).

All patients were followed for 45 days from admission. Mortality status was determined through hospital medical records and verified by the national electronic health information system. Multivariable statistical modeling will be applied to adjust for baseline clinical and radiological variables.

This study aims to provide new insights into the potential role of spleen dynamics as a prognostic biomarker in acute ICH, supporting early risk stratification strategies in the neurocritical care setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Radiologically confirmed diagnosis of intraparenchymal intracerebral hemorrhage (ICH)
* Underwent baseline and 72-hour follow-up brain CT scans
* Underwent abdominal ultrasound at baseline
* Provided written informed consent prior to participation

Exclusion Criteria:

* Incomplete or missing imaging data (brain CT or abdominal ultrasound)
* Loss to follow-up or withdrawal of consent before 45 days post-discharge
* Presence of conditions known to cause splenomegaly (e.g., hematological malignancies, liver cirrhosis, infectious diseases)
* Age under 18 years
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 42 adult patients (≥18 years) diagnosed with intraparenchymal intracerebral hemorrhage confirmed by radiological imaging. Eligible patients underwent both baseline and 72-hour follow-up brain CT scans and abdominal ultrasound. Participants were consecutively enrolled from those presenting to the Emergency Department. Patients with incomplete imaging data, loss to follow-up before 45 days post-discharge, or conditions causing splenomegaly were excluded. Informed consent was obtained from all participants.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in spleen volume (ΔSpleen) from baseline to 72 hours | Baseline (within 24 hours of admission) and 72 hours
  Spleen volume will be measured using abdominal ultrasound volumetry at baseline and at 72 hours. Change (ΔSpleen) will be calculated as the difference between baseline and 72-hour measurement.
  Unit of Measure: milliliters (mL)

SECONDARY OUTCOMES:
45-day all-cause mortality | 45 days
  Mortality status will be assessed through hospital records and the national electronic health system.
  Unit of Measure: percentage of patients (%)
Change in hematoma volume (ΔHematoma) from baseline to 72 hours | Hematoma volume change calculated as 72-hour minus baseline measurements
  Hematoma volume will be measured using brain CT volumetry at baseline and at 72 hours. Change (ΔHematoma) will be calculated as the difference between baseline and 72-hour measurement.
  Unit of Measure: milliliters (mL)
Baseline Glasgow Coma Scale (GCS) scores | Baseline Glasgow Coma Scale measured within 24 hours of admission
  The Glasgow Coma Scale (GCS) is a standardized neurological scale used to assess the level of consciousness in patients with acute brain injury. It ranges from 3 (deep coma or death) to 15 (fully awake and oriented). In this study, baseline GCS scores are recorded upon patient admission, within 24 hours of spontaneous intracerebral hemorrhage diagnosis. The score is derived from three components: eye opening, verbal response, and motor response, each rated on a numerical scale and summed to provide the total GCS score. This measure serves as an objective indicator of initial neurological status.

CONTACTS AND LOCATIONS:
Overall Officials: Cagdas Yildirim, Assistant Professor, Principal Investigator — Ankara City Hospital Bilkent; Kadir Yenal, Attending Physician, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Emergency Medicine Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared include anonymized demographic information (age, sex), clinical characteristics (baseline and 72-hour brain CT findings, abdominal ultrasound results), treatment details, and 45-day follow-up outcomes (survival status). All shared data will be fully de-identified to protect patient privacy. The dataset will exclude any direct identifiers such as names, addresses, or personal identification numbers. Data sharing will support secondary analyses and meta-analyses related to intracerebral hemorrhage and spleen volume without compromising confidentiality. Access will be granted upon reasonable request and after approval by the study's data sharing committee.
Supporting Information: Study Protocol, SAP
Time Frame: The individual participant data (IPD) and supporting documentation will be available starting six months after the publication of the primary study results. Data access will remain open for a period of five years from the start date. During this time, qualified researchers can request access to the de-identified dataset and associated metadata for secondary analyses. After the five-year period, data availability will be reviewed and may be extended depending on data management policies and resource availability.
Access Criteria: Access to the individual participant data (IPD) and supporting documentation will be granted to qualified researchers who submit a formal data request outlining the objectives and methods of their proposed analysis. Researchers must agree to use the data solely for approved research purposes and to maintain confidentiality and data security. The shared data will include fully de-identified participant information and relevant metadata necessary to understand the dataset. Access will be provided through a secure data sharing platform or via direct transfer after approval by the study's data sharing committee. Requests will be reviewed based on scientific merit and ethical considerations.